CLINICAL TRIAL: NCT01366235
Title: Clinical Trial for Evaluation of Ethnic Differences in Pharmacokinetics of Chloroquine, an Anti-malarial Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-0214
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — chloroquine diphosphate

ARMS (4):
- Southeast Asians (Experimental)
  Interventions: Drug: chloroquine phosphate 1000 mg
- Korean (Experimental)
  Interventions: Drug: chloroquine phosphate 1000 mg
- Caucasians (Experimental)
  Interventions: Drug: chloroquine phosphate 1000 mg
- Africans (Experimental)
  Interventions: Drug: chloroquine phosphate 1000 mg

INTERVENTIONS:
Drug: chloroquine phosphate 1000 mg — 1000 mg, 1day

SUMMARY:
Chloroquine is an anti-malaria agent. This study is designed to evaluate inter-ethnic differences of therapeutic effect of chloroquine and search the cause of these ethnic differences. For this purpose, chloroquine will be administered to four ethic groups of Korean, Caucasian, African and Southeast Asian and chloroquine concentration in blood will be measured. The result of this study will be helpful in finding more adequate dosing regimen of chloroquine in patients with malaria.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 - 50 male subjects (6 Koreans, 6 Caucasians, 6 Africans and 6 Southeast Asians)
* Subjects with body weight ≥ 45 kg and within ±20% of the ideal body weight : Ideal body weight = (height [cm] - 100)x0.9.

Exclusion Criteria:

* Subjects who have drunken habitually (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the study period from 2 days prior to the first administration of investigational product and during this study.
* Subjects deemed ineligible by investigator based on other reasons, including abnormal laboratory values or diseases.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic evaluation | within 30 days
  maximum of concentration(Cmax)

SECONDARY OUTCOMES:
pharmacokinetic evaluations | within 30 days
  Area under the time-concentration curve(AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr